CLINICAL TRIAL: NCT01651507
Title: Evaluation of Outcome of Adult Pulmonary Langerhans Cell Histiocytosis Based on Lung HRCT and Lung Function. A Multicenter Retrospective Study
Brief Title: Evaluation of Outcome of Adult Pulmonary Langerhans Cell Histiocytosis Based on Lung HRCT and Lung Function
Acronym: HLP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HLP
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2010-09

CONDITIONS: Pulmonary Langerhans Cell Histiocytosis
Keywords: Pulmonary Langerhans cell histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HLP: Patients with pulmonary LCH from eight teaching hospitals evaluated between June 1989 and February 2005 were considered for this study, if they were followed for at least 6 months and evaluated by ≥ 2 lung HRCT and lung function tests at the same time or within a 2 months period

SUMMARY:
this is a multicenter retrospective study on patients with pulmonary LCH who were sequentially evaluated by concomitant lung HRCT and lung function testing. The objectives of this study were: 1) to determine the changes over time of lung function parameters in patients with pulmonary LCH; 2) to compare the variations of HRCT and lung function results during follow-up; 3) to address the respective interest of these investigations for identifying the patients who eventually will experience a progression of their disease.

DETAILED DESCRIPTION:
Pulmonary Langerhans cell histiocytosis (pulmonary LCH) is an uncommon disorder, characterized by the accumulation of CD1a+ Langerhans cells (LCs) organized in granulomas that develop in, and destroy the wall of distal bronchioles. In adults the disease occurs predominantly in young smokers from both genders, with a peak incidence at 20-40 yrs of age, although female may be slightly older. High resolution computed tomography (HRCT) of the lung has provided a considerable input for the diagnosis of pulmonary LCH.

We conducted a multicenter retrospective study on patients with pulmonary LCH who were sequentially evaluated by concomitant lung HRCT and lung function testing. The objectives of this study were: 1) to determine the changes over time of lung function parameters in patients with pulmonary LCH; 2) to compare the variations of HRCT and lung function results during follow-up; 3) to address the respective interest of these investigations for identifying the patients who eventually will experience a progression of their disease. Results of this study may help to improve the management of patients with adult pulmonary LCH.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary HLP diagnosed between June 1989 and February 2005

Exclusion Criteria:

* followed up for less than 6 months
* with less than 2 lung HRCT and lung function tests at the same time or within a 2 month period

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with pulmonary LCH
  * enrolled in eight teaching hospitals
  * evaluated between June 1989 and February 2005
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 1989-06; Primary Completion 2005-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Impairment of lung function | 5 years
  a decrease ≥10% of FEV1 or FVC, or decrease ≥15% of DLCO. Conversely, if the FEV1or FVC increased of ≥10%, or DLCO ≥15%
obstructive pattern | 5 years
  FEV1/FVC ratio <70%
restrictive pattern | 5 years
  TLC <80% of predicted value
lung HRCT cystic score | 5 years
  The extent of cystic lesions (including thick- and thin- walled cysts) was assessed for each of the 6 defined lung areas on HRCT and classified as follows: 0 (no cyst); 1 (<25%); 2 (25-49%); 3 (50-75%) and 4 (>75%) of the lung surface analyzed. For the whole lung, the maximal value for cystic HRCT score was of 24

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, Paris, France

REFERENCES:
- [Result] Tazi A, Marc K, Dominique S, de Bazelaire C, Crestani B, Chinet T, Israel-Biet D, Cadranel J, Frija J, Lorillon G, Valeyre D, Chevret S. Serial computed tomography and lung function testing in pulmonary Langerhans' cell histiocytosis. Eur Respir J. 2012 Oct;40(4):905-12. doi: 10.1183/09031936.00210711. Epub 2012 Mar 22. PMID 22441752